CLINICAL TRIAL: NCT03812900
Title: Comparative, Conceptual, Randomized Clinical Study to Investigate Superiority of Newly Developed Over Basic Echinacea Formulations for the Treatment of Acute Symptoms of Respiratory Tract Infections
Brief Title: Superiority of Newly Developed Over Basic Echinacea Formulations for the Treatment of Respiratory Tract Infections
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: A. Vogel AG (Industry)
Collaborators: Cantonal Hospital of St. Gallen (Other); Labormedizinisches Zentrum Dr. Risch (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5'000'155
Record Dates: First submitted 2018-09-07; First posted 2019-01-23 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Formulation A (Experimental): Echinacea purpurea alcoholic extract lozenges (novel formulation)
  Interventions: Drug: Echinacea purpurea alcoholic extract
- Formulation B (Experimental): Echinacea purpurea alcoholic extract spray (novel formulation)
  Interventions: Drug: Echinacea purpurea alcoholic extract
- Formulation C (Active Comparator): Echinacea purpurea alcoholic extract tablet (basic formulation, reference)
  Interventions: Drug: Echinacea purpurea alcoholic extract
- Formulation D (Active Comparator): Echinacea purpurea alcoholic extract, drops (basic formulation, reference)
  Interventions: Drug: Echinacea purpurea alcoholic extract

INTERVENTIONS:
Drug: Echinacea purpurea alcoholic extract — Different galenic forms with Echinacea purpurea alcoholic extract from herb and roots (95:5%)

SUMMARY:
This is a comparative, conceptual, randomized clinical study to investigate newly developed over basic Echinacea formulations for the treatment of acute symptoms of respiratory tract infections. 400 adults will be recruited, of which approximately 300 will develop a common cold or a influenza-like infection. Two newly developed and two existing Echinacea formulations (solid/liquid) will be randomly dispensed at inclusion for treatment of maximal 3 infections. Treatment starts at first signs of infection and lasts for a maximum of 10 days or until symptom resolution. Nasopharynx samples will be collected for analysis of common viral respiratory agents throughout treatment. Safety and efficacy variables will be assessed.

DETAILED DESCRIPTION:
The monocentre trial compares two newly developed pharmaceutical forms of Echinacea (extract from Echinacea purpurea Herba and Radix; lozenges or spray) with two basic and authorised pharmaceutical forms (tablets or drops; comparator groups) for the treatment of acute symptoms of the common cold and/or influenza-like illness (ILI) in adults. Trial subjects are preventatively screened and included in the study (n = 400). If they show acute symptoms of a common cold or ILI during the study period, they are instructed to call the study centre to have confirmed the indication for treatment and begin with the treatment, they are randomized to (1:1:1:1 randomization into one of four groups). The primary endpoint is the time until remission of respiratory symptoms with the new pharmaceutical forms compared to the basic forms during the first episode. Secondary endpoints include remission of all treated episodes (max. 3 episodes), remission times comparison between different pharmaceutical forms (e.g. lozenges vs. spray, lozenges vs. drops etc), reduction of viral load on day 5 and 9 compared to day 1 of treatment (nasopharyngeal swabs), differences in safety (blood parameters before and during treatment), differences in number of adverse events, tolerance and efficacy assessed by the patients.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Signed Informed Consent

Exclusion Criteria:

* Younger than 18 years
* Participation in another clinical study in the past 30 days
* Permanent intake of antimicrobial, antiviral, immune suppressive substances
* Surgical intervention in the 3 months prior to inclusion or planned surgery during period of observation
* Known diabetes melitus
* Known and treated atopy or asthma bronchiale
* Cystic fibrosis, bronchopulmonale dysplasia, COPD
* Known diseases of the immune system, degenerative illnesses (e.g. auto-immune disorders like AIDS or leukemia, myeloma)
* Known metabolic or resorptive disorders
* Known chronic liver diseases (chronic hepatitis, liver cirrhosis)
* Known chronic kidney insufficiency
* Serious health issues (reduced health status, autoimmune illness, tumorous illness)
* Known allergy to plants of compositae family (camomille, dandelion) or to any substances of the investigational product
* At inclusion known pregnancy or planned pregnancy during period of investigation (required: active contraception for women of childbearing year)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Time to remission from initial episodes | maximally 10 days
  duration until respiratory symptoms are solved

SECONDARY OUTCOMES:
Time to remission from overall episodes | maximally 10 days
  duration until respiratory symptoms are solved
Cross-comparison of remissions between formulations | maximally 10 days
  duration until respiratory symptoms are solved
Development of single respiratory symptoms | maximally 10 days
  Comparison of respiratory symptom scores between formulations, adapted Jackson Score [0-3, 0=absent, 3=severe]
Development of respiratory symptom sum score | maximally 10 days
  Comparison of symptom sum scores between formulations, adapted Jackson Score [0-27, each 0=absent, 3=severe]
Absence from School/Work | during acute respiratory episodes, 7 days each
  Number of days absent from work or school
Reduction of viral load in nasopharyngeal samples | day 1, day 5, day 9
  Comparison of virus titer at day 5 and 9 i.c. to day 1
Subjective assessment of efficacy by patient | At end of treatment cycle of 10 days
  Comparisons of subjective efficacy assessments between patients [0=poor; 1=moderate; 2=good; 3=very good]. Inofficial scale and and global method of assessing patients satisfaction re efficacy.
Blood safety (red and white cell count) | At Inclusion visit and day 5 of infection
  Change of blood parameters before (V1) and after treatment (V2)
Blood safety (creatinin [umol/l]) | At Inclusion visit and day 5 of infection
  Change of blood parameters before (V1) and after treatment (V2)
Blood safety (ALT [ukat/l]) | At Inclusion visit and day 5 of infection
  Change of blood parameters before (V1) and after treatment (V2)
Blood safety (AST [ukat/l]) | At Inclusion visit and day 5 of infection
  Change of blood parameters before (V1) and after treatment (V2)
Blood safety (Bilirubin [umol/l]) | At Inclusion visit and day 5 of infection
  Change of blood parameters before (V1) and after treatment (V2)
Acceptance of treatment | At end of treatment cycle of 10 days
  Question:"would you use the medicament again?"
Concomitant medication and -therapy | during acute respiratory episodes of 10 days
  Incidence of concomitant medication and -therapy
adverse events | during acute respiratory episodes, from day 1 until follow up at day 17 - 21
  occurrence of adverse events during treatment with Echinacea
Subjective assessment of tolerability by patient | At day 10 of every treatment cycle
  Comparisons of subjective tolerability assessments between patients [0=poor; 1=moderate; 2=good; 3=very good]. Inofficial scale and and global method of assessing patients satisfaction re tolerability.

CONTACTS AND LOCATIONS:
Locations (1):
- Cantonal Hospital St. Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sumer J, Keckeis K, Scanferla G, Frischknecht M, Notter J, Steffen A, Kohler P, Schmid P, Roth B, Wissel K, Vernazza P, Klein P, Schoop R, Albrich WC. Novel Echinacea formulations for the treatment of acute respiratory tract infections in adults-A randomized blinded controlled trial. Front Med (Lausanne). 2023 Apr 17;10:948787. doi: 10.3389/fmed.2023.948787. eCollection 2023. PMID 37138742